CLINICAL TRIAL: NCT05344456
Title: Switching PVC Response ''Atrial Pace'' in ST JUDE Medical or Abbott ICD (Implantable Cardioverter Defibrillator) or CRT-D (Cardiac Resynchronization Therapy) Devices to Off Mode Decreases the Burden of Atrial Tachycardia
Brief Title: PVC Response ''Atrial Pace'' Inducing Atrial Tachycardias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Markus Sane, M.D, PhD, Cardiologist, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/627/2022
Record Dates: First submitted 2022-04-14; First posted 2022-04-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Tachycardia
Keywords: premature ventricular complex; pacemaker; arrythmia
MeSH Terms: conditions — Ventricular Premature Complexes; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVC response ''Off'' (Experimental)
  Interventions: Device: Change in the device PVC algorithm to ''Off''

INTERVENTIONS:
Device: Change in the device PVC algorithm to ''Off'' — PVC algorithm change from Atrial Pace mode to Off

SUMMARY:
Premature ventricular contractions (PVC) are common phenomenon and occasionally retrograde conduction from ventricle to atrium occurs and may cause pacemaker mediated tachycardia. In response certain Abbott (former St Jude Medical) pacemakers have a specific PVC response algorithm ''Atrial Pace''. In this algorithm the PVARP (Post Ventricular Atrial Refractory Period) is extended to 480ms but the initial 150ms of the PVARP is deemed absolute. If atrial sensed event occurs after absolute PVARP the PVARP terminates and atrial pace follows after 330ms alert period. Two case reports exists where patients atrial tachycardia were suspected to be induced by this algorithm. In Helsinki University Hospital an index patient with multiple atrial tachycardia episodes was recognized in late 2020 where the cause of the tachycardias was suspected to be the PVC response algorithm ''Atrial Pace''. After programming the algorithm from Atrial Pace to off mode the patient had none atrial tachycardias during 2021. After investigating all the patients with physiological ICD (Implantable Cardioverter Defibrillator) or CRT-D (Cardiac Resynchronization Therapy) device and analyzing remote monitoring transmissions from the year 2020 we found 25 patients with similar atrial tachycardia episodes possibly induced by the PVC response ''Atrial Pace''.

DETAILED DESCRIPTION:
The device of the subjects participating to the study is interrogated and the PVC response algorithm is switched from ''Atrial Pace'' to ''Off'' mode.

Subjects are also requested to fulfill the EQ-5D-3L and ICD8 questionaries before the change in the device programming and after the 12 months surveillance.

ELIGIBILITY:
Inclusion Criteria:

* ST Jude Medical or Abbott physiological ICD or CRT-D device
* PVC response setting ''Atrial Pace''
* Atrial tachycardia episode duration > 30s preceded by ventricular extrasystole and atrial pace in year 2020 or 2021

Exclusion Criteria:

* Permanent atrial fibrillation, duration ≥ 6 months before the enrollment to the study
* PVC response has been switched off before enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Number of atrial tachycardia episodes per participant which is initiated after PVC followed by atrial sensed event and atrial pace after 330ms delay. | The number of these episodes is compared between year 2020 and 12 months preceding the change in the programming setting and 12 months afterwards.
  Atrial tachycardia episode is considered as an episode which duration is >30s and atrial rate > 180 beats per minute.
Number of any atrial tachycardia episodes and overall duration of atrial tachycardia episodes per participant. | The number of these episodes and overall duration of all atrial tachycardia episodes is compared between year 2020 and 12 months preceding the change in the programming setting and 12 months afterwards.
  Atrial tachycardia episode is considered as an episode which duration is >30s and atrial rate > 180 beats per minute.

SECONDARY OUTCOMES:
Composite Change in the quality of life analyzed with EQ-5D-3L and ICD8 questionaries'. | baseline and after 12 months surveillance
  In EQ-5D-3L questionary the quality of life is measured in scale from 0 to 100 and in ICD8 questionary in scale from 0 to 32. The overall score in both of the questionaries is compared at two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Sane, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman DJ, Chasten T, Anderson K, Mullenix J, Rider K, Sun AY. Premature ventricular contraction response-induced new-onset atrial fibrillation. HeartRhythm Case Rep. 2018 Nov 30;5(3):120-123. doi: 10.1016/j.hrcr.2018.11.012. eCollection 2019 Mar. No abstract available. PMID 30891406
- [Background] Liu Y, Yuan X. Logic Analysis of Arrhythmia Triggered by Pacemaker Special Functions - An Educational Presentation. Braz J Cardiovasc Surg. 2021 Jun 1;36(3):412-415. doi: 10.21470/1678-9741-2020-0630. PMID 34387977